CLINICAL TRIAL: NCT06990828
Title: The Effect of Frenkel's Stabilization Exercises on Balance, Physical Performance, and Fear of Falling in Geriatric Individuals
Brief Title: Frenkel Exercises in Geriatric Balance and Fall Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Assos. Prof, Okan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29.09.2021/142
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Healthy Aging
Keywords: balance; fear of falling; physical performance; frenkel stabilitation exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): Participants included in the study will undergo a program of Frenkel Stabilization Exercises.
  Interventions: Other: Frenkel Stabilization Exercises

INTERVENTIONS:
Other: Frenkel Stabilization Exercises — Participants included in the study will undergo a program of Frenkel Stabilization Exercises.

SUMMARY:
Aging is a natural process starting from birth and progressing through childhood and adulthood, marked by physical and mental decline, including musculoskeletal, cognitive, and motor deterioration. It often results in common conditions such as visual and hearing impairments, sleep disturbances, urinary incontinence, hypertension, dementia, cardiovascular diseases, osteoarthritis, osteoporosis, gait abnormalities, and frequent falls. Osteoporosis contributes to decreased bone density and structural integrity, impairing posture and balance.

Balance, maintained through the integration of vestibular, visual, and proprioceptive inputs, becomes impaired with aging, increasing fall risk and injury. Falls are a major cause of morbidity and mortality in the elderly, affecting one-third of individuals over 65 annually. Risk factors are classified as intrinsic (e.g., muscle weakness, gait issues, chronic diseases) and extrinsic (e.g., poor lighting, unsafe flooring).

Physical inactivity in older adults leads to reduced strength, endurance, flexibility, and overall functional health, requiring greater effort for daily tasks. Early detection of reduced physical fitness and the implementation of targeted exercise programs are essential to prevent functional decline and falls. Evidence supports the effectiveness of strength and balance exercises in reducing fall-related injuries and fear of falling.

Exercise improves both physical and psychological well-being in older adults, enhancing social participation, flexibility, strength, bone mineral density, and spinal mobility. This study aims to investigate the effects of Frenkel's Stabilization Exercises on balance, physical performance, and fear of falling in healthy geriatric individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 years and older,
* Individuals who are able to comprehend the questions in the data collection forms,
* Volunteers who are willing to participate in the study.

Exclusion Criteria:

* Individuals with painful or painless orthopedic conditions that could significantly affect physical performance,
* Individuals with serious orthopedic or systemic disorders that would prevent them from participating in exercise.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Tinetti Balance and Gait Test | 20 days
  This test evaluates balance ability and walking under two main categories. The first nine items assess balance, while the following seven items evaluate gait.
  The total score of the balance items gives the balance score, and the total of the gait items gives the gait score.
  The sum of both scores represents the overall test score. Higher scores indicate a lower risk of falling.
The Alusti Test | 20 days
  The physical performance of the participants will be assessed using the Alusti Test.
  This test, designed for geriatric individuals, consists of 10 items and is scored out of 100 to evaluate physical performance.
  According to the total score, levels of mobility are classified as follows:
  0-30: Completely dependent mobility 31-40: Severely dependent mobility 41-50: Moderately dependent mobility 51-60: Mildly dependent mobility 61-75: Good mobility 76-90: Very good mobility 91-100: Excellent mobility
The International Fall Efficacy Scale | 20 days
  The International Fall Efficacy Scale (FES-I) will be used to assess fear of falling.
  The scale evaluates older adults' confidence and level of fear of falling during activities of daily living.
  It has been translated into many languages and is widely used. The total score ranges from 16 to 64, with higher scores indicating a greater fear of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided